CLINICAL TRIAL: NCT04656665
Title: The Effectiveness of Low-dose Aspirin on Preventing Pre-eclampsia in High-risks Pregnant Women
Brief Title: The Effectiveness of Aspirin on Preventing Pre-eclampsia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ThirdGuangzhouMU
Record Dates: First submitted 2020-11-11; First posted 2020-12-07 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Pre-Eclampsia
Keywords: Pre-eclampsia, Aspirin
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 75mg (Experimental): Take 75mg of aspirin daily in tihis group
  Interventions: Drug: Aspirin
- 100mg (Active Comparator): Take 100mg of aspirin daily in this group
  Interventions: Drug: Aspirin
- blank (No Intervention): Not taking aspirin in this group

INTERVENTIONS:
Drug: Aspirin — For patients at high risk of pre-eclampsia, start taking aspirin from 12-20 weeks of pregnancy
  Other Names: Acetylsalicylic acid
  Arms: 100mg; 75mg

SUMMARY:
This study will explore the effectiveness of low-dose aspirin on preventing pre-eclampsia in high-risks pregnant women by comparing the incidence of pre-eclampsia and pregnancy outcomes.

DETAILED DESCRIPTION:
Currently，low-dose aspirin is a commonly used drug to prevent pre-eclampsia. Many guidelines recommend starting low-dose aspirin in early pregnancy in high-risks pregnant women. However, the applicable population and use method of aspirin are still controversial in clinical practice. This study will explore the effectiveness and use method of low-dose aspirin by comparing the incidence of pre-eclampsia and pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55 years
* Gestational age between 12-20 weeks of pregnancy
* High risk of developing pre-eclampsia

  * At least one of the following risk factors: Pre-eclampsia in a previous pregnancy , Multiple pregnancy，Diabetes Mellitus(Type 1 or 2), Chronic Hypertension，Renal disease, Autoimmune disease.
  * At least two of the following risk factors: Primiparity，Pre-pregnancy Body Mass Index ≥28kg/m2, Age ≥35 years, Family members have a history of pre-eclampsia.
* Maternal informed conset obtained

Exclusion Criteria:

* Contraindication to aspirin therapy (including but not limited to allergy and high bleeding risk)
* Patient with known intention to terminate pregnancy
* Fetal abnormalities detected （including but not limited to major fetal malformation and FGR）
* Severe heart, liver, renal disease who can not burden the experiment
* Alcohol and drug abuse
* Being in another drug experiment within 3 months

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2022-12-14 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of pre-eclampsia | 1 year
  Record the number of pre-eclampsia in each group and compare whether there are statistical differences in the incidence of each group

SECONDARY OUTCOMES:
Preterm birth | 1 year
  Record the number of preterm in each group and compare whether there are statistical differences in the incidence of each group
Fetal growth restriction | 1 year
  Record the number of FGR in each group and compare whether there are statistical differences in the incidence of each group
Placental abruption 4/5000 Placental abruption | 1 year
  Record the number of placental abruption in each group and compare whether there are statistical differences in the incidence of each group
Postpartum hemorrhage | 1 year
  Record the number of postpartum hemorrhage in each group and compare whether there are statistical differences in the incidence of each group